CLINICAL TRIAL: NCT06634121
Title: Efficacy of Mitraclip Vs. PASCAL for the Treatment of Mitral Regurgitation in an All-comer Population
Acronym: LEAFLET I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Jörg Hausleiter, Deputy chief, LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEAFLET I
Record Dates: First submitted 2024-08-26; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Mitral Regurgitation; Valvular Heart Disease; Heart Failure
Keywords: Mitral Regurgitation; TEER; MitraClip; PASCAL
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Valve Diseases; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MitraClip (Active Comparator)
  Interventions: Device: Transcatheter mitral valve edge-to-edge repair (M-TEER)
- PASCAL (Active Comparator)
  Interventions: Device: Transcatheter mitral valve edge-to-edge repair (M-TEER)

INTERVENTIONS:
Device: Transcatheter mitral valve edge-to-edge repair (M-TEER) — M-TEER is performed via a transfemoral venous approach. After puncture of the interatrial septum the mitral valve is repaired using either the PASCAL or MitraClip device.

SUMMARY:
To investigate potential differences in procedural outcomes of both commercially available transcatheter edge-to-edge mitral valve repair devices in a non-selected clinical setting.

DETAILED DESCRIPTION:
In the context of M-TEER, two different systems (MitraClip vs. PASCAL) are CE certified and clinically available. In the case of non-complex anatomy, both systems are comparable in terms of effectiveness. Whether this holds true in cases of complex or highly complex anatomy in an "Allcomer patient population" is currently unclear.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or above 18 years
* Written consent
* Heart Team recommends M-TEER

Exclusion Criteria:

* Mitral Stenosis (MV mean PG > 5 mmHg)
* Cardiogenic shock or hemodynamic instability at the time of intervention
* Active endocarditis
* Participant in another interventional cardiology study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Postprocedural residual MR measured by 3D EROA | During the index procedure
  residual MR measured by 3D EROA as continuous parameter

SECONDARY OUTCOMES:
Reduction in MR EROA | During the index procedure
  Reduction in MR EROA from baseline to postprocedural (relative and absolut value)
Comparing EROA in complex vs. non-complex patients | During the index procedure
  Evaluation according to EROA reduction
Postprocedural MV opening area | During the index procedure
  Postprocedural MV opening area (planimetric)
Postprocedural MV inflow gradient | During the index procedure
  Mean pressure gradient and pressure halftime
SLDA | During the index procedure, at 30-day follow-up and at 1-year follow-up
  Single Leaflet Device Attachment
Conversion to surgery or re-imaging of the MV | During the index procedure, at 30-day follow-up and at 1-year follow-up
  Conversion to surgery (urgently or elective) or re-imaging of the MV
Stratification by MR etiology | During the index procedure, at 30-day follow-up and at 1-year follow-up
  Primary vs. Secondary MR
Combined endpoint of mortality, repeat MV intervention or HHF | During the index procedure, at 30-day follow-up and at 1-year follow-up
  Assessed at 30-days and 1-year
Quality of Life | At 30-day follow-up and at 1-year follow-up
  Measured using the KCCQ Score
Exertional dyspnea | At 30-day follow-up and at 1-year follow-up
  NYHA functional class

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Hausleiter, Prof. Dr., Principal Investigator — LMU Klinikum; Ludwig Weckbach, PD Dr., Principal Investigator — LMU Klinikum
Locations (1):
- LMU Klinikum, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided